CLINICAL TRIAL: NCT03531268
Title: Prospective Study to Evaluate the Clinical Utility of Perioperative Pharmacogenomic Testing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Need improve the strategy
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CQuentia NGS, LLC (Unknown)
Responsible Party: Principal Investigator, Srdjan Nedeljkovic, Anesthesiologist, Associate Professor of Anaesthesia, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2018P000454
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Pharmacogenomic Analysis; Clinical Utility; Outcomes
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: All subjects meeting inclusion/exclusion criteria will undergo pharmacogenomic testing. The group for which testing is thought to have clinical utility will be compared to the group for which testing is thought to have no clinical utility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGx testing has clinical utility (Active Comparator): These are subjects whose PGx testing is judged to have clinical utility and whose clinical care may be modified. Modifications may include altering doses or types of drugs given based on metabolic profile of the patient.
  Interventions: Other: PGx Testing
- PGx testing has no clinical utility (No Intervention): These are subjects whose PGx testing is judged to have no clinical utility. Care "as usual" is provided, and there are no changes in drug selection or dosing based on the results of PGx testing.

INTERVENTIONS:
Other: PGx Testing — Pharmacogenomic (PGx) testing will be administered to all subjects. The results of PGx testing will be evaluated for clinical utility. Subjects will be evaluated based on whether PGx testing has clinical utility or has no clinical utility.
  Arms: PGx testing has clinical utility

SUMMARY:
In the perioperative realm, studies have demonstrated an association of genotype with efficacy of medications applicable to the surgical setting. A clinical association exists between the genotype of various genes and with opioid efficacy and toxicity - specifically for drugs such as oxycodone, codeine, morphine, fentanyl, and tramadol. More studies are needed to assess the effects of personalized dosing of analgesics during the perioperative process for various surgical procedures. The application of Pharmacogenomic testing (PGx) to perioperative medicine is novel, has much potential for growth and may potentially improve outcomes. However, successful implementation of a system to evaluate PGx and integrate results into clinical decision-making is challenging and has not been adequately assessed. The investigators propose to conduct PGx testing for patients undergoing surgery, evaluate its clinical utility, and assess outcomes. The investigators hypothesize that PGx testing may ultimately lead to a decrease in adverse events and improved outcomes in the perioperative period.

DETAILED DESCRIPTION:
Potential subjects will participate in screening with a minimum of 4 days prior to their planned surgery. The study involves obtaining mouth swab samples for genetic testing and employing standardized measures for PGx testing of subjects preoperatively.

Study staff will pre-screen potential subjects scheduled at the preoperative center or on surgeons' operative schedules. The study team member will ask the treating clinician involved with the care of a patient for permission to speak to the patient. The physician or a member of the research staff will describe the study to potentially eligible patients and a study investigator will obtain consent. After meeting inclusion and exclusion criteria, subjects who agree to participate in the study will complete study questionnaires and provide a swab sample for PGx analysis.

Trained members of the research staff will obtain a buccal swab sample from each subject who has given informed consent to participate in study procedures. The buccal swab will be packaged and shipped to an outside laboratory for processing and the conduct of the PGx testing. The results of the PGx testing will be provided in a standardized report and sent back to the research staff conducting the study. Typically, the turn-around for shipping the sample and obtaining the results will be 4 days. The results will be available to the anesthesiologist prior to the patient's surgery.

Prior to the initiation of the scheduled surgery, the anesthesiologist will be asked to complete a questionnaire about the clinical utility of PGx testing for that subject. In the perioperative group of subjects for whom clinicians find clinical utility for PGx testing (experimental group), outcomes will be compared to the remaining subjects (control group) for whom PGx testing was felt not to have any clinical utility.

After surgery, there will be two assessment periods. Clinical outcomes and the quality of the subject's recovery from surgery will be assessed postoperatively at 24 hours +/-4 hours after surgery by directly interviewing each study subject and reviewing the electronic medical record. Additional assessments of subjects will be conducted by review of the electronic medical record at 30 days +/- 3 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older at screening.
2. Adults with qualifying insurance coverage.
3. Subjects scheduled to undergo elective surgery with an expected hospitalization 24 hrs =/- 4 hrs after surgery.
4. American Society of Anesthesiology (ASA) physical status 1, 2, or 3.
5. One or more of the following:

   * Subjects prescribed 4 or more medications at time of surgery.
   * Any subject prescribed any one of the following medication categories: opioid, benzodiazepine, antidepressant, antipsychotic, stimulant, mood stabilizer, NSAIDs, anti-epileptic drugs.
   * Any subject prescribed any one of the following medication categories: antiplatelet therapy, anticoagulant drugs.
6. Able to provide informed consent, adhere to the study protocol, and complete all study assessments.

Exclusion Criteria:

1. Subjects who do not have insurance coverage for PGx testing.
2. Subjects who are expected to have surgery prior to the ability to obtain the results of the pharmacogenomic testing (generally it takes 4 days to obtain the results of testing).
3. Subjects who are not being prescribed 4 or more medications, or who are not receiving any of the medication categories noted in the inclusion criteria.
4. Planned multiple surgical procedures within the 30-day study follow up period.
5. Clinically significant medical or psychiatric disease that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other disease that would cause the subject to be unable to comply with the study requirements.
6. Administration of an investigational drug within 30 days prior to providing PGx testing, or planned administration of an investigational product during the subject's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Clinical Utility | The day of surgery or the day prior
  The anesthesiologist will be shown the results of PGx testing and will complete a "Clinical Utility Questionnaire" regarding the clinical utility of PGx testing for the subject. The responses will be rated: 0 = no utility; 1 = some utility; 2 = significant utility. The larger value (2) is considered as having a higher utility for this scale.

SECONDARY OUTCOMES:
Intraoperative and postoperative use of opioids | 24 hrs +/- 4 hrs after surgery
  The use of intraoperative and postoperative use of opioids will be measured (morphine mg equivalents)
Duration times (surgery, anesthesia, length of stay in PACU) | 24 hrs +/- 4 hrs after surgery
  Surgical duration and anesthesia duration times, length of stay in PACU (duration will be measured in minutes)
Pain Assessment | 24 hrs +/- 4 hrs after surgery
  Pain Numeric Rating Scale, 0 - 10 (0 = no pain, 10 = maximum pain) (lower values = better outcome)
Postoperative Nausea and Vomiting | 24 hrs +/- 4 hrs after surgery
  Postoperative Nausea and Vomiting Scale (0 = no nausea/vomiting, 200 = maximal nausea/vomiting) (lower values = better outcome)
Sedation and Delirium Assessment | 24 hrs +/- 4 hrs after surgery
  Richmond Agitation and Sedation Scale (-5 = unarousable, 0 = alert and calm, +4 = combative) (values = 0 are best outcome)
Subject Satisfaction | 24 hrs +/- 4 hrs after surgery
  Subject Satisfaction Questionnaire (1 = extremely dissatisfied, 5 = extremely satisfied) (higher values = best outcome)
Quality of Recovery | 24 hrs +/- 4 hrs after surgery
  Quality of Recovery Questionnaire (0 = poor, 150 = excellent) (higher values = best outcome)
Length of stay in hospital after surgery | 30 days
  Length of stay in the hospital after surgery (days)(lower number = best outcome)
Opioid Prescriptions | 30 days
  Amount of opioids prescribed after surgery (morphine mg equivalents) (lower amount = best outcome)
Hospital Readmissions | 30 days
  Number of times readmitted to hospital within 30 days after surgery (lower number = best outcome)
Emergency Room Visits | 30 days
  Number of emergency room visits within 30 days after surgery (lower number = best outcome)
Unscheduled Phone Calls | 30 days
  Number of unscheduled phone calls to the doctor's office within 30 days after surgery (lower number = best outcome)
Unscheduled Office Visits | 30 days
  Number of unscheduled visits to the doctor's office within 30 days after surgery (lower number = best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan S Nedeljkovic, MD, Study Director — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cregg R, Russo G, Gubbay A, Branford R, Sato H. Pharmacogenetics of analgesic drugs. Br J Pain. 2013 Nov;7(4):189-208. doi: 10.1177/2049463713507439. PMID 26516523
- [Background] Jannetto PJ, Bratanow NC. Utilization of pharmacogenomics and therapeutic drug monitoring for opioid pain management. Pharmacogenomics. 2009 Jul;10(7):1157-67. doi: 10.2217/pgs.09.64. PMID 19604091